CLINICAL TRIAL: NCT02741297
Title: A Multi-Center Controlled Study to Characterize the Real-world Outcomes of High Rate Spinal Cord Stimulation Therapy Using Boston Scientific (BSC) PRECISION Spinal Cord Stimulator System
Brief Title: VELOCITY: A Study to Characterize Real-World Outcomes of Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91113648
Record Dates: First submitted 2016-04-14; First posted 2016-04-18 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Cord Stimulation (SCS) System (Experimental): Boston Scientific (BSC) PRECISION SCS System with MultiWave Technology
  Interventions: Device: Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) System — Boston Scientific (BSC) PRECISION SCS System with MultiWave Technology

SUMMARY:
The primary objective of this study is to characterize the real-world outcomes of spinal cord stimulation (SCS) therapy as an aid in the management of chronic intractable pain of the trunk, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable low back pain using the Boston Scientific (BSC) PRECISION Spinal Cord Stimulator System with MultiWave Technology.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the real-world outcomes of spinal cord stimulation (SCS) therapy as an aid in the management of chronic intractable pain of the trunk, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable low back pain using the Boston Scientific (BSC) PRECISION Spinal Cord Stimulator System with MultiWave Technology.

ELIGIBILITY:
Key Inclusion Criteria:

* Complaint of persistent or recurrent low back pain for at least 180 days prior to Screening
* Willing and able to comply with all protocol-required procedures and assessments/evaluations
* Subject signed a valid, ethics committee (EC)-approved informed consent form (ICF) provided in local language

Key Exclusion Criteria:

* High surgical risk
* Previous spinal cord stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)
* A female who is pregnant, is breastfeeding, or is of childbearing potential and planning to get pregnant during the course of the study or not using adequate contraception.
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study
* Any diagnosis or condition that, in the clinician's best judgment, might confound reporting of study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, Principal Investigator — St Bartholomew's Hospital, London, UK
Locations (5):
- Schreiber Klinik, München, Germany
- Azienda Ospedale Monaldi, Naples, Italy
- Ziekenhuis Rijnstate, Velp, Netherlands
- United Kingdom (2):
  - Southmead Hospital Bristol, Bristol
  - St. Bartholomews Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Cord Stimulation (SCS) System
Started | 73
Completed | 59
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation (SCS) System
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Average Low Back Pain Scores (NRS) [Mean (Standard Deviation); unit: units on a scale] — Average low back pain will be based on the 0-10 Numerical Pain Rating Scale (NRS) where 0 indicates no pain and 10 is worst pain (higher scores indicate more pain)
  units on a scale | 7.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Low Back Pain Responders
Description: Percentage of low back pain responders at 3 months post-activation with no increase in opioids from Baseline to 3 months post-activation
Time Frame: 3 months
Population: For " All subjects without outlier sites", data for those sites with outlier subjects were removed.
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation (SCS) System
Number analyzed (Participants) | 59
Participants
  All Subjects | 25
  All subjects without outliers: number analyzed (Participants) | 41
  All subjects without outliers | 23

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Spinal Cord Stimulation (SCS) System
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 6/73
Other Adverse Events (participants affected / at risk) | 4/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (SCS) System (N=73)
Angina Unstable (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Circulatory Collapse (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (SCS) System (N=73)
Implant Site Infection (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02741297/Prot_SAP_000.pdf